CLINICAL TRIAL: NCT05144048
Title: Outpatient Induction of Labor With Oral Misoprostol: A Multicenter Randomized-controlled Trial
Brief Title: Outpatient Induction of Labor With Oral Misoprostol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); Nordlandssykehuset HF (Other); Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 261787/2021
Record Dates: First submitted 2021-11-03; First posted 2021-12-03 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2022-09

CONDITIONS: Induction of Labor
Keywords: induction; outpatient; misoprostol; childbirth experience

STUDY DESIGN:
Intervention Model Description: All eligible women will be recruited form a midwife and/or doctor. After the inclusion the women will be randomized to either inpatient or outpatient setting.
Masking Description: The women will be randomized using a secure survey tool to an inpatient or outpatient setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction of labour with oral misoprostol, inpatient setting (Active Comparator): These women receive all treatment in the maternity unit.
  Interventions: Other: Inpatient setting
- Induction of labour with oral misoprostol, outpatient setting (Experimental): These women are observed 2 hours after they receive one dose of oral misoprostol before they leave the maternity unit.
  Interventions: Other: Outpatient setting

INTERVENTIONS:
Other: Inpatient setting — These women stay at the maternity unit
  Arms: Induction of labour with oral misoprostol, inpatient setting
Other: Outpatient setting — These women leave the maternity unit
  Arms: Induction of labour with oral misoprostol, outpatient setting

SUMMARY:
Induction of labor is an increasingly used intervention in obstetrics due to expanding indications, which more often includes relatively healthy women with uncomplicated pregnancies. While induction of labor traditionally is offered in an inpatient setting, a shift towards an outpatient setting is increasing despite insufficient evidence regarding safety and effectiveness. Oral misoprostol is easy for the pregnant women to administer and the risk of uterine hyperstimulation with fetal heart rate changes is found to be low. Strong evidence concludes that oral misoprostol is preferable as an induction agent and is recommended by the World Health Organization (WHO).

The investigators will perform a multicenter randomized-controlled trial comparing labor induction in an outpatient versus inpatient setting, aiming to increase knowledge on outpatient induction of labor with oral misoprostol. The study is based on experiences and findings from a recently performed pilot trial and targets a large group of relatively healthy pregnant women where induction of labor is decided.

The investigators hypothesize that women induced in an outpatient setting will be more satisfied than women induced in an inpatient setting.

DETAILED DESCRIPTION:
After induction of labor is decided the women will be recruited according to inclusion and exclusion criteria's.

The inpatient induction group will receive the following treatment:

Oral misoprostol 25ug every two hours and a cardiotocography for fetal monitoring every 4-6 hours until start of contractions, the next 48 hours while admitted to the maternity ward. The participating women will be transferred to the labor ward by start of contractions or need for closer fetal surveillance and/or analgesia.

The outpatient induction group will receive the following treatment:

These participating women receive the first oral misoprostol 25ug at the maternity unit. After two hours if the cardiotocograph is normal and there are no signs of contractions, these women go home. At home, the women will continue to take 25ug misoprostol every two hours until 22 pm or until the contractions begin. Maximum time spent at home is 48 hours and maximum number of tablets is 12 during this period (6 tablets each day). The women will also receive oral and written information regarding when to return to the maternity ward. Information sheets for the midwives and included women will be adapted from those used in the pilot study.

If the contractions are still absent after 48 hours or a maximum of 12 tablets (6 per day), all women (both inpatient and outpatient) are admitted to the maternity ward for further induction of labor. All women will receive equal standard of care including fetal surveillance after admittance to the hospital. Further follow up is in accordance with standard procedure of the maternity ward. Questions about fidelity to the proposed protocol across sites will be asked in the patient questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 37 gestational weeks, vertex presentation, single pregnancy
* Age ≥ 18 years
* Understand and read Norwegian
* Distance to hospital less than 1 hour
* Normal ultrasound including:

  * fetal movements
  * amniotic fluid (deepest single vertical pocket) > 2 cm
  * estimated fetal weight ≥ -15% (≥ 10 percentile)
* Normal antenatal cardiotocography
* Women with stable hypertension and uncomplicated preeclampsia without indication for inpatient treatment can be included after individual assessment.
* Access to partner or contact person at home for transportation to hospital

Exclusion Criteria:

* Premature rupture of membranes
* Uterine scar
* BMI ≥ 40
* Abnormal fetal Doppler (if examined); umbilical artery pulsatility index ≥ 95 percentile and/or cerebroplacental ratio <1
* Fetal anomaly or chromosomic / genetic disorder
* Grand multipara (P≥4)
* Cognitive barriers
* Pregnancy complications such as preeclampsia requiring in-hospital treatment, insulin dependent diabetes or other conditions associated with risk of fetal hypoxia during labor
* Signs of infection or serious health problems
* Favorable cervix and / or previous obstetric history providing contraindications for induction with misoprostol
* Combined risk factors, individually evaluated by the attending obstetrician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Maternal childbirth experience and maternal experience with induction of labor | up to 12 days after delivery
  The women will answer electronic questionaires at inclusion and postpartum

SECONDARY OUTCOMES:
Labor outcomes | From 1 hour to average of 48 hours
  Hours from start induction and start active labor
Cost per delivery | through study completion, an average of 1 year
  We will calculate the differences of costs and effects of one or more alternatives, and present the differences in the form of a ratio (ICER), i.e. the cost per unit of health outcome or effect. We will calculate cost-effectiveness (δ costs / δ effects) to evaluate whether outpatient induction shows to be dominant strategy regarding patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Janne Rossen, MD, PhD, Principal Investigator — Sorlandet HF
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset HF, Bodø
  - Østfold Hospital Trust, Fredrikstad
  - Sorlandet Hospital Trust, Kristiansand
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO recommendations: Induction of labour at or beyond term. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK535795/ PMID 30629393
- [Background] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803
- [Background] Alfirevic Z, Aflaifel N, Weeks A. Oral misoprostol for induction of labour. Cochrane Database Syst Rev. 2014 Jun 13;2014(6):CD001338. doi: 10.1002/14651858.CD001338.pub3. PMID 24924489
- [Background] McDonagh M, Skelly AC, Tilden E, Brodt ED, Dana T, Hart E, Kantner SN, Fu R, Hermesch AC. Outpatient Cervical Ripening: A Systematic Review and Meta-analysis. Obstet Gynecol. 2021 Jun 1;137(6):1091-1101. doi: 10.1097/AOG.0000000000004382. PMID 33752219
- [Background] Helmig RB, Hvidman LE. An audit of oral administration of Angusta(R) (misoprostol) 25 microg for induction of labor in 976 consecutive women with a singleton pregnancy in a university hospital in Denmark. Acta Obstet Gynecol Scand. 2020 Oct;99(10):1396-1402. doi: 10.1111/aogs.13876. Epub 2020 May 19. PMID 32311758
- [Background] Ten Eikelder ML, Oude Rengerink K, Jozwiak M, de Leeuw JW, de Graaf IM, van Pampus MG, Holswilder M, Oudijk MA, van Baaren GJ, Pernet PJ, Bax C, van Unnik GA, Martens G, Porath M, van Vliet H, Rijnders RJ, Feitsma AH, Roumen FJ, van Loon AJ, Versendaal H, Weinans MJ, Woiski M, van Beek E, Hermsen B, Mol BW, Bloemenkamp KW. Induction of labour at term with oral misoprostol versus a Foley catheter (PROBAAT-II): a multicentre randomised controlled non-inferiority trial. Lancet. 2016 Apr 16;387(10028):1619-28. doi: 10.1016/S0140-6736(16)00084-2. Epub 2016 Feb 3. PMID 26850983
- [Derived] Austad FE, Kessler J, Magnussen EB, Pripp AH, Rossen J. Outpatient Versus Inpatient Induction of Labour With Oral Misoprostol: A Multicentre Randomised-Controlled Trial. BJOG. 2025 Oct;132(11):1562-1573. doi: 10.1111/1471-0528.18296. Epub 2025 Jul 24. PMID 40704452